CLINICAL TRIAL: NCT05519982
Title: Sleep Treatment Education Program (STEP-1): An Online Educational Intervention for Insomnia in Cancer Survivors
Brief Title: Sleep Treatment Education Program-1 (STEP-1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Recklitis, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-516; 1R21CA267857 (NIH)
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivors; Insomnia
Keywords: Cancer Survivors; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Treatment Education Program (STEP-1) (Experimental): Prior to being randomized, all participants will complete health questionnaires.
  Participants assigned to the Sleep Treatment Education Program (STEP-1) group will receive online instruction on making changes to sleep habits and health behaviors.
  Participants will be contacted at 1 month and 2 months after the education session to complete follow up online questionnaires.
  Interventions: Behavioral: Sleep Treatment Education Program (STEP-1)
- Enhanced Usual Care: Relaxation Education (Active Comparator): Prior to being randomized, all participants will complete health questionnaires.
  Participants assigned to the Enhanced Usual Care group will receive information on relaxation techniques to improve sleep
  Participants will be contacted at 1 month and 2 months after the education session to complete follow up online questionnaires.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Sleep Treatment Education Program (STEP-1) — Video conference instruction on behavioral changes to improve sleep.
  Arms: Sleep Treatment Education Program (STEP-1)
Behavioral: Enhanced Usual Care — Video conference instruction on relaxation techniques to improve sleep.
  Arms: Enhanced Usual Care: Relaxation Education

SUMMARY:
The purpose of the study is to learn if single session online education programs can help improve cancer survivors' sleep.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of cancer survivors with clinically significant symptoms of insomnia to evaluate the efficacy of the cognitive-behavioral intervention Sleep Treatment Education Program-1 (STEP-1).

Participants in this study will be randomized to either the behavioral education session, Sleep Treatment Education Program-1 (STEP-1), which will instruct them on how to make changes to their sleep habits and behaviors or an enhanced usual care control program which will provides them with access to online relaxation programs and instruct them about how these programs can help improve sleep.

Participation in the study involves:

* Taking part in a 60-90 minute, one-on-one session using the Zoom video conference platform and completing a brief online questionnaires.
* Completing an approximately 10 minute follow-up questionnaire online with a brief phone call 4, and 8 weeks after the education session. An additional optional insomnia questionnaire will be requested at one month after the 8 week follow-up.
* Participants will receive a $25 gift card upon completing 4 & 8 week questionnaires.

It expected that about 70 people will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-89
* History of a cancer diagnosis (except non-melanoma skin cancer) ≥ 1 year prior
* No active cancer therapy (excluding chemoprevention) in the past four months, and no further therapy planned
* Significant insomnia as evidenced by an Insomnia Severity Index score ≥12
* Regular access to the internet on a daily basis
* Able to read and write in English

Exclusion Criteria:

* Survivors who report ever being diagnosed with Bipolar Disorder.
* Survivors who report ever being diagnosed with a Seizure Disorder or have experienced a seizure in the past 12 months.
* Intention to adjust (decrease or increase) use of any prescribed or over-the-counter medications taken to decrease insomnia during the study period.
* Survivors diagnosed with sleep apnea who have declined treatment or are not adherent with treatment (as assessed by screening questions, see Appendix A).
* Survivors with suspected sleep apnea who have not completed an evaluation by a sleep specialist (as assessed by screening questions, see Appendix A).
* Usual bedtime does not fall between 5:00 pm and 5:00 am.
* Employment that involves irregular sleep patterns, such as shift-work or frequent long-distance travel across time zones, or employment in a position that could impact public safety (such as air traffic-controller, operating heavy machinery)
* Any impairment (e.g., hearing, visual, cognitive) that interferes with the ability to complete all study procedures independently.
* Prior participation in a research study which provided an educational or behavioral intervention for insomnia.
* Prior participation in a behavioral treatment or patient education program for insomnia delivered at the Dana-Farber Cancer Institute, or at Boston Children's Hospital.
* Participation in behavioral or educational interventions for insomnia in the 2 years prior to enrollment. This includes in-person as well as synchronous and asynchronous online insomnia programs, but not independent use of books, workbooks or other written self-help materials addressing insomnia.

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Recklitis, PhD, MPH, Principal Investigator — Dana-Farber Cancer Insitute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Bice BL, Michaud AL, McCormick KG, Miklos EM, Descombes ID, Medeiros-Nancarrow C, Zhou ES, Recklitis CJ. Sleep Treatment Education Program for Cancer Survivors: Protocol for an Efficacy Trial. JMIR Res Protoc. 2024 Nov 28;13:e60762. doi: 10.2196/60762. PMID 39608001

RESULTS

PARTICIPANT FLOW:
Groups:
- STEP-1: Participants received a single 75-minute synchronous videoconference intervention session based on cognitive behavioral therapy components of sleep hygiene, stimulus control, and cognitive restructuring
- Relaxation (Control): Participants received a single 60-minute synchronous videoconference education session based on relaxation exercises such as progressive muscle relaxation, paced breathing, and guided imagery
Period: Intervention Session and Evaluation
Arm/Group | STEP-1 | Relaxation (Control)
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0
Period: Required Follow-up
Arm/Group | STEP-1 | Relaxation (Control)
Started | 35 | 35
Completed | 34 | 33
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0
Period: Optional Extended Follow-up
Arm/Group | STEP-1 | Relaxation (Control)
Started | 33 | 32
Completed | 24 | 20
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 9 | 12

BASELINE CHARACTERISTICS:
Population: From the original 70 participants who began the study and completed the Baseline questionnaire, two participants were lost to follow-up and one withdrew following the education session (reflected in the Participant Flow chart). Those three participants were not included in the analyzed sample reported here (n=67).
Groups:
- Total: Total of all reporting groups
Arm/Group | STEP-1 | Relaxation (Control) | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (10.7) | 60.8 (11.9) | 61.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 31 | 31 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 1 | 1
Insomnia Severity Index [Mean (Standard Deviation); unit: Units on a scale] — The Insomnia Severity Index (ISI) is a 7-item measure used to evaluate insomnia severity (e.g. dissatisfaction with sleep and worry about sleep problems). Item response values are totaled to calculate a total ISI score ranging from 0-28, with higher scores indicating more insomnia symptom burden.
  Units on a scale | 15.8 (3.0) | 15.5 (3.8) | 15.8 (3.3)
Profile of Mood States - Short Form (Total Mood Disturbance) [Mean (Standard Deviation); unit: Units on a scale] — The Profile of Mood States-Short Form (POMS-SF) is a 35-item measure of mood. Item responses are totaled to calculate scores on 7 subscales. The Total Mood Disturbance (TMD) score used in the study is calculated by adding together the scores of 5 subscales, Anger-Hostility, Confusion-Bewilderment, Depression-Dejection, Fatigue-Inertia, Tension-Anxiety, then subtracting the score from the Vigor-Activity subscale. TMD scores range from -20 to 100 higher scores indicating greater impairment.
  Units on a scale | 9.7 (14.1) | 13.6 (19.4) | 11.7 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Change at 8 Weeks
Description: The Insomnia Severity Index (ISI) is a 7-item measure used to evaluate insomnia severity (e.g. dissatisfaction with sleep and worry about sleep problems). Item response values are totaled to calculate a total ISI score ranging from 0-28, with higher scores indicating more insomnia symptom burden.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | STEP-1 | Relaxation (Control)
Number analyzed (Participants) | 34 | 33
Units on a scale | 7.3 (4.2) | 9.5 (4.6)

2. Secondary Outcome: Profile of Mood States Change at 8 Weeks
Description: The Profile of Mood States-Short Form (POMS-SF) is a 35-item measure of mood. Items responses are totaled to calculate scores on 7 subscales: Anger-Hostility, Confusion-Bewilderment, Depression-Dejection, Fatigue-Inertia, Tension-Anxiety, Vigor-Activity, and Friendliness. The Total Mood Disturbance (TMD) score used in the study is calculated by adding together the scores of 5 subscales, Anger-Hostility, Confusion-Bewilderment, Depression-Dejection, Fatigue-Inertia, Tension-Anxiety, then subtracting the score from the Vigor-Activity subscale. TMD scores range from -20 to 100 with higher scores indicating greater impairment.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | STEP-1 | Relaxation (Control)
Number analyzed (Participants) | 34 | 33
Units on a scale | .85 (11.7) | 4.2 (13.6)

3. Secondary Outcome: Profile of Mood States Change at 4 Weeks
Description: as for outcome 2
Time Frame: Baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | STEP-1 | Relaxation (Control)
Number analyzed (Participants) | 34 | 33
Units on a scale | 3.4 (14.9) | 6.4 (15.4)

4. Secondary Outcome: Change in Sleep Quality
Description: The PROMIS Sleep Disturbance Short Form 8b (PROMIS-SD) is an 8 item scale used to assess sleep disturbances and their impact on overall sleep quality. Items include specific sleep problems (e.g., restless sleep) as well as satisfaction with sleep quality and amount of sleep. Item responses are summed to calculate a Total score, with raw scores (range 8-40) translated into t-scores (mean = 50, SD= 10). Higher PROMIS-SD Total t-scores indicate greater levels of sleep disturbance.
Time Frame: Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | STEP-1 | Relaxation (Control)
Number analyzed (Participants) | 34 | 33
Units on a scale | 52.2 (4.3) | 53.1 (4.6)

5. Secondary Outcome: Sleep Duration
Description: Total sleep time in hours per night calculated from the Consensus Sleep Diary-Morning
Time Frame: Administered at 8 week follow-up
Measure: Median (Inter-Quartile Range); unit: Time (in hours per night)
Arm/Group | STEP-1 | Relaxation (Control)
Number analyzed (Participants) | 34 | 33
Time (in hours per night) | 7.0 [6.3 to 7.9] | 7.3 [6.2 to 7.9]

6. Secondary Outcome: Insomnia Severity Change at 4 Weeks
Description: as for outcome 1
Time Frame: Baseline to 4 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | STEP-1 | Relaxation (Control)
Number analyzed (Participants) | 34 | 33
Units on a scale | 8.6 (4.4) | 11.7 (3.3)

7. Other Pre Specified Outcome: Intervention Session Usability & Satisfaction
Description: Study specific participant checklist describing ease of use, acceptability and credibility of intervention
Time Frame: Up to 4 weeks post-intervention
Reporting Status: Not Posted, anticipated posting 2026-07

8. Other Pre Specified Outcome: Intervention Satisfaction Summary
Description: Brief participant questionnaire to provide feedback about the intervention and how it could be improved.
Time Frame: Completed at the 8-week post-intervention timepoint
Reporting Status: Not Posted, anticipated posting 2026-07

9. Other Pre Specified Outcome: Coaching Satisfaction Summary
Description: Brief participant questionnaire to provide feedback about coaching session. could be improved.
Time Frame: Up to 13 weeks post-intervention
Reporting Status: Not Posted, anticipated posting 2026-07

10. Other Pre Specified Outcome: Insomnia Symptoms at 16 Weeks (Optional)
Description: After completing 8-week follow-up, participants will be asked if they are willing to complete one additional Insomnia Severity Scale 8 weeks later.
Time Frame: At 16 weeks post-intervention
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: From enrollment to 8 weeks for all participants, additional follow-up to 12 weeks for participants in optional coaching session
Description: This was a minimal risk educational intervention. Participants self-report on significant health changes in their own words.
Arm/Group | STEP-1 | Relaxation (Control)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT05519982/Prot_SAP_000.pdf